CLINICAL TRIAL: NCT04914286
Title: A Multi-center, Single-arm, and Open-label Phase Ib/II Study Exploring the Safety/Tolerability, Pharmacokinetics, and Efficacy of GFH018 in Combination With Toripalimab in the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Study of GFH018 in Combination With Toripalimab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH018X0201
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GFH018+Toripalimab (Experimental): Patient will be dosed in GFH018 in combination with Toripalimab. In the PhaseIb part, the dose levels will be escalated following the Bayesian optimal interval (BOIN) design. In the Phase II part, patients will be assigned based on tumor type(s).
  Interventions: Drug: GFH018; Drug: Toripalimab

INTERVENTIONS:
Drug: GFH018 — Subjects are planned to be dosed in oral GFH018 tablets twice daily for a continuous 14 days in a 28 days cycle (7days on 7days off may be tested based on available data from phase I dose escalation study of single agent). the starting dose of GFH018 will be derived from the maximum safe dose explored in rom phase I dose escalation study of single agent.
Drug: Toripalimab — Subjects are planned to be dosed at 3 mg/kg Toripalimab as an intravenous infusion once every 2 weeks.

SUMMARY:
The purpose of the study is to evaluate the safety/tolerability, pharmacokinetics, and preliminary efficacy of GFH018 in combination with Toripalimab in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumors, progressed on at least first line therapy.
2. Has sufficient organ functions.
3. Eastern Cooperative Oncology Group Performance Status (ECOG P.S.) ≤ 1. Subject with tumor involvement of the liver must have the Child-Pugh score of 0-7.
4. Life expectancy≥12 weeks.
5. Female or male subjects of child-bearing potential must agree to use effective contraceptive methods from the signing of the informed consent to 90 days after the last administration of the study drug. Fertile female subjects must have negative pregnancy test results within 7 days (inclusive) before administration.

In addition, eligible patients in phase II part must meet the following criteria:

1. Histologically or cytologically confirmed diagnosis of unresectable or metastatic advanced tumors of specific types: hepatocellular carcinoma, cholangiocarcinoma/gallbladder cancer (except carcinoma of ampulla), pancreatic cancer, colorectal cancer, urothelium carcinoma, cervical cancer, head and neck squamous cell carcinoma, esophageal cancer and nasopharyngeal carcinoma.
2. At least one measurable lesion (according to RECIST 1.1).

Exclusion Criteria:

1. Impaired cardiac function or clinically significant cardiac diseases.
2. With acute or chronic infections.
3. With active central nervous system metastases, including symptomatic brain metastases, meningeal metastases, spinal cord compression, or requiring treatment with glucocorticoids, antiepileptic drugs, anticonvulsant drugs, or mannitol.
4. With known active autoimmune diseases or a history of autoimmune diseases within 1 year prior to enrollment.
5. With clinically significant gastrointestinal diseases.
6. Uncontrollable or symptomatic ascites, pleural effusion or pericardial effusion.
7. With previous or present interstitial pneumonia.
8. With other uncontrolled systemic diseases, such as hypertension and diabetes.
9. Diagnosed with other malignant tumors within 3 years prior to starting study drug, except for cured carcinoma in situ of cervix and skin basal cell carcinoma.
10. With diseases requiring immunosuppressant therapy, or requiring prednisone > 10 mg/day or equivalent dose of similar drugs during the study period.
11. Subjects who have been treated with immunosuppressant drugs within 28 days prior to starting study drug, except for topical and inhaled cortisol and systemic cortisol of physiological dose (prednisone < 10 mg/day or equivalent dose of similar drugs).
12. Subjects who have received live vaccine, attenuated vaccine within 28 days prior to starting study drug, or plans to receive live vaccine, attenuated vaccine during treatment or within 30 days after the last administration.
13. Subjects who have been treated with radiotherapy, chemotherapy, targeted therapy, endocrine therapy, immunotherapy, and other anti-tumor therapies, or other investigational drugs within 5 half-life periods or within 28 days (whichever is shorter) prior to starting study drug.
14. Subject who has received major surgeries (except for needle biopsy) that may affect the administration or study evaluation within 28 days prior to starting study drug.
15. Subjects who have received strong inhibitor or inducer of CYP3A4, or herbal medicine/traditional Chinese medicines within 5 half-life periods or within 2 weeks (whichever is shorter) prior to starting study drug.
16. Subjects who have received combined treatment of drugs targeting TGF-β and PD-(L)1, including combination of antibody and small molecule or bispecific antibody.
17. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Phase Ib：Incidence of dose-limiting toxicity (DLT) events | 28 days
Phase II: ORR (Objective Response Rate) | approximately 6 months after first dose

CONTACTS AND LOCATIONS:
Locations (3):
- Linear Clinical Research Ltd, Perth, Western Australia, Australia
- China (2):
  - Sun Yat-sen university cancer center, Guangzhou, Guangdong
  - Shang hai east hospital, Shanghai, Shanghai Municipality

DOCUMENTS (1):
  • Study Protocol (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT04914286/Prot_000.pdf